CLINICAL TRIAL: NCT04435847
Title: Phase 1b, Double-Blind, Placebo-controlled Study of Safety and Efficacy of HST 001 in Male Subjects With Male Pattern Hair Loss
Brief Title: Safety and Efficacy of HST 001 in Male Pattern Hair Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Histogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HST 001-AES-003-HG
Record Dates: First submitted 2020-05-26; First posted 2020-06-17 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2020-08

CONDITIONS: Male Pattern Hair Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HST 001 (Experimental): HST 001 (also known as hair stimulating complex [HSC]) is a mixture of growth factors secreted by human dermal fibroblasts when cultured in proprietary bioreactors which are then harvested and concentrated to specific ranges.
  Interventions: Biological: HST 001
- Placebo - Phosphate Buffered Saline (Placebo Comparator): Phosphate Buffered Saline
  Interventions: Other: Phosphate Buffered Saline

INTERVENTIONS:
Biological: HST 001 — Participants will receive intradermal injections at 3 timepoints only: week 0, week 6 and week 12. At each of these 3 interventional visits they will receive 0.1 mL X 20 injections spaced approximately 0.8 - 1.2 cm apart from one another of active treatment (HST 001).
  Arms: HST 001
Other: Phosphate Buffered Saline — Participants will receive intradermal injections at 3 timepoints only: week 0, week 6 and week 12. At each of these 3 interventional visits they will receive 0.1 mL X 20 injections spaced approximately 0.8 - 1.2 cm apart from one another of placebo control (Phosphate Buffered Saline).
  Arms: Placebo - Phosphate Buffered Saline

SUMMARY:
HST 001 (also known as hair stimulating complex [HSC]) is a mixture of growth factors secreted by human dermal fibroblasts when cultured in proprietary bioreactors which are then harvested and concentrated to specific ranges. In both preclinical studies and in previous clinical trials, HSC has been shown to be safe, with no serious adverse events reported. This protocol design is based on the completed Phase 1 study in women which used a similar investigational product (Study 16-HIS002-US; HSC660), and includes specific objective efficacy endpoints (macrophotography) to measure Target Area Hair Counts (TAHC) after three separate doses of product separated by six weeks (week 0, week 6, week 12) and comparing to placebo treated group

DETAILED DESCRIPTION:
* Single center, randomized, controlled, parallel-design study in participants with mild to moderate hair loss on a Norwood-Hamilton (N-H) Scale
* Double-blind: Evaluating Investigator (EI) and participants are blinded; Treating Investigator (TI) is not blinded
* Investigational product is randomly assigned to subjects upon enrollment and will receive either HST 001 or placebo (phosphate buffered saline [PBS]). Injections will be delivered via 1 mL syringes with 31 Gauge needles to the target depth of 1.75 mm, using a slow injection technique and holding the needle in position for count of 3-4 seconds. Each injection will provide 0.1 mL and a total of 20 injections will be given in the scalp with particular attention to the leading edge of the vertex and the temporal recession areas
* Participants will receive intradermal injections at 3 timepoints only: week 0, week 6 and week 12. At each of these 3 interventional visits they will receive 0.1 mL X 20 injections spaced approximately 0.8 - 1.2 cm apart from one another. Dosing will be split between the leading edge of the vertex region (~10 injections covering 10.18 cm2) and in each temporal recession area (~5 injections covering 7.07cm2) in each.
* Adverse Events (AEs) will be monitored to ensure safety of participants throughout the study
* Efficacy will be assessed at Week 18 and Week 26 via macrophotography and TAHC by the Canfield HairMetrix System

ELIGIBILITY:
Inclusion Criteria

1. Must be 25 to 55 years of age inclusive, at the time of signing the informed consent
2. Should be in good general health with a healthy scalp with no cutaneous disorder determined by medical history or physical examination
3. Are classified as III Vertex (3 Vertex), IV (4) and V (5) under the N H Classification for male pattern hair loss (MPHL). Subjects should have some thinning in both the vertex and temporal regions of the scalp
4. Willing to maintain the same hair-style during the study period. No razor shaving of head (bald) prior to study start and throughout the study period
5. Must be Male.
6. Willing to have two dot tattoos of the scalp
7. Willing to have an approximately 1.0 cm2 area of hairs clipped in the vertex region and 0.5 cm2 in one temporal recession area at each visit where macrophotography is conducted
8. Willing to comply with scheduled 7 visits in 26 weeks (or screening in + 6 = 7 visits)
9. Willing to continue normal hair care shampoo throughout the course of the study
10. Willing to maintain the same hair care routine and forgo the use of new scalp products, throughout the study
11. Willing to undergo routine venipuncture for safety laboratory testing as well as a blood spot test for Vitamin D level analysis
12. Capable of giving informed consent
13. Fluent and literate in English
14. Able to follow instructions and likely to complete all study visits as assessed by investigator and staff

Exclusion Criteria

1. History of keloid formation or significant hyperpigmentation
2. History of other forms of hair loss - Alopecia areata, trichotillomania, scarring alopecia etc.
3. History of acute or chronic illness that in the opinion of the investigator might confound the results of the study including some drug medications
4. Active skin diseases (eczema, atopic dermatitis, psoriasis, skin cancer, sun-damaged skin with actinic keratosis on the scalp, etc.) in or around the area to be treated
5. Routine use of prescription anti inflammatory medications, immunosuppressive drugs, or antihistamine medications
6. Use of topical drugs or other cosmetics on the scalp
7. Use of over the counter (OTC) or prescriptive topical hair treatments, including hair transplantation during the last 6 months
8. Currently using a hair system or wig
9. History of hair transplants or scalp reduction surgery
10. History of allergy or intolerance to lidocaine and/or epinephrine
11. Use of hair dye within 3 days of the treatments, otherwise, willing to maintain the same hair color for the study duration
12. Current enrollment in an investigational drug or device study
13. Has tattoos or scars in scalp that would interfere with visual assessment
14. Is an employee of the investigator's site, and employee or representative of Histogen, investor, or a relative with one of the above
15. Has a condition or is in a situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with participant's involvement in the study
16. Known allergy to rice
17. Known allergy to bovine products

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Participant assessment of procedural pain. | 26 Weeks
  Participant assessment of procedural pain as captured on the "Subject Self Assessment Questionnaire for Pain." Minimum score is 1, Maximum score is 5, higher score means worse outcome.
Participant assessment of pain or other treatment site responses. | 26 Weeks
  Participant assessment of pain or other treatment site responses as captured on "Subject Self Assessment Questionnaire for Pain." The number and percent of participants reporting each sensation will be collected.
Adverse Events | 26 Weeks
  Safety and tolerability of HST 001 by comparing adverse events to baseline
Serum collection for Anti-Drug Antibodies | 26 Weeks
  Serum collection for testing for Anti-Drug Antibodies
Absolute change from baseline total hairs in the target area (TAHC) of the vertex. | 18 Weeks
  Absolute change from baseline total hairs in the target area (TAHC) of the vertexes measured by Canfield's HairMetrix macrophotography system at week 18 compared to week 0 (Baseline).

SECONDARY OUTCOMES:
Absolute change from baseline total TAHC of the right temporal region. | 18 Weeks
  Absolute change from baseline total TAHC of the right temporal region as measured by Canfield's HairMetrix macrophotography system at week 18 compared to week 0 (Baseline).
Absolute change from baseline total TAHC in the vertex and right temporal areas. | 26 Weeks
  Absolute change from baseline total TAHC in the vertex and right temporal areas as measured by Canfield's HairMetrix macrophotography system at week 26 compared to week 0 (baseline).
Absolute change from baseline in non-vellus and vellus hair count in the vertex and right temporal area. | 26 Weeks
  Absolute change from baseline in non-vellus and vellus hair count in the vertex and right temporal area as measured by Canfield's HairMetrix macrophotography system at week 18 compared to week 0; and week 26 compared to week 0.
Cumulative thickness density (total hair count x total hair width) in the vertex and temporal areas. | 26 Weeks
  Cumulative thickness density (total hair count x total hair width) in the vertex and temporal areas derived from Canfield's HairMetrix system measurements at week 18 and week 26.
Percent change from baseline in TAHC, non-vellus hair counts, vellus hair counts at the vertex and right temporal areas. | 26 Weeks
  Percent change from baseline in TAHC, non-vellus hair counts, vellus hair counts at the vertex and right temporal areas (separately) comparing week 0 to week 18 and week 0 to week 26.
Participant global assessment of hair growth. | 26 Weeks
  Participant global assessment of hair growth from global photos on the "Subject Self Assessment Questionnaire for Efficacy," patient reported outcome measure for hair growth. Minimum score is 7 and Maximum score is 35. Lower scores indicate a better outcome.
Evaluating investigator global assessment of hair growth. | 26 Weeks
  Evaluating investigator global assessment of hair growth from global photos, captured on the "Global Assessment Likert scale for Hair Growth ." Minimum score is -3 and Maximum score is +3. Positive scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- California Dermatology & Clinical Research Institute, Encinitas, California, United States